CLINICAL TRIAL: NCT06438536
Title: STEPS (Social Cognitive Training Enhancing Pro-functional Skills): A Clinical Randomized Trial Evaluating the Effect of a Virtual Reality-based Intervention for Adults With Autism.
Brief Title: STEPS: A Virtual Reality-based Intervention for Adults With Autism.
Acronym: STEPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Principal Investigator, Louise Birkedal Glenthoej, DMSc, PhD, psychologist with specialization in psychiatry and specialist in psychotherapy, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-23055504
Record Dates: First submitted 2024-05-23; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Autism Spectrum Disorder
Keywords: Randomized clinical trial (RCT); Virtual Reality (VR); Social cognitive training; Cognitive remediation; Digital intervention
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: The study is a high-quality randomized, assessor-blinded parallel-groups superiority clinical trial fulfilling the CONSORT criteria for non-pharmacological treatment. A total of 140 adults with ASD will be allocated to receive either 12 weeks of Virtual Reality-based Social Cognitive Training (VRSCT) + treatment as usual (TAU) or TAU. All participants will be assessed at baseline and at 3- and 6-months post-baseline.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Stratified block randomization with concealed randomization sequences will be conducted after baseline assessment. Independent assessors blinded to the treatment will evaluate outcomes. Analysis of outcomes will be carried out following the intention-to-treat principles.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality-based Social Cognitive Training (VRSCT) (Experimental): Patients in the experimental group will be offered 10 individual sessions of targeted, virtual reality assisted psychotherapy embedded in cognitive behavioral therapy (CBT), that aims at enhancing social cognition and daily life functioning. If the patient consents, two additional sessions will be offered in which the patient's relatives are invited to participate (one in the beginning of treatment and one at the end of treatment). The aim of the relative involvement is to enhance transfer from the therapy to the patients daily life. The treatment will be conducted by psychologists with an extensive knowledge in providing virtual reality assisted therapy. The treatment is manualized, and the therapists will receive ongoing supervision by a senior clinician having ≥ 25 years of experience in conducting assessment, treatment, and research with the autism spectrum population.
  Interventions: Behavioral: Virtual Reality-based Social Cognitive Training
- Treatment as Usual (TAU) (No Intervention): The treatment-as-usual (TAU) group will receive the standard treatment offered to adults diagnosed with ASD in Denmark. This commonly consists of four psychoeducational sessions as well as limited supportive counseling. Some adults with ASD also receive practical help in daily life situations in community settings. The TAU will be mapped upon trial completion.

INTERVENTIONS:
Behavioral: Virtual Reality-based Social Cognitive Training — Virtual reality assisted social cognitive training embedded in cognitive behavioral therapy, that aims at enhancing social cognition and daily life functioning.
  Arms: Virtual Reality-based Social Cognitive Training (VRSCT)

SUMMARY:
The goal of this clinical trial is to learn if a new Virtual Reality-based intervention will be effective in treating social cognitive challenges in adults with autism.

The main questions it aims to answer are:

1. Is Virtual Reality-based social cognitive training effective in reducing social cognitive deficits and improving psychosocial functioning, quality of life, and clinical symptoms in adults with ASD?
2. Is Virtual Reality-based social cognitive training cost-effective?

Researchers will compare Virtual Reality-based pro-functional, Social Cognitive Training (VRSCT) to treatment as usual (TAU) to evaluate effectiveness.

Participants will be allocated to receive either VRSCT once a week in addition to treatment as usual (TAU) or TAU alone for 3 months. All participants will undergo a thorough assessment at baseline, and at 3 and 6 months post-baseline.

DETAILED DESCRIPTION:
Adults with autism spectrum disorders (ASD) constitute an increasingly recognized population with largely unaddressed public health needs. Research on effective interventions for adults with ASD lags far behind that dedicated to children with ASD, as well as other psychiatric disorders.

Adults with ASD show prominent social cognitive deficits that impede their daily functioning such as being able to interact socially, to achieve adequate vocational functioning (i.e. job/educational achievements) as well as inflicting immensely on their quality of life. At current, no robust and replicated evidence exists on a pro-functional treatment targeting social cognitive deficits in adults with ASD.

Virtual reality-based treatment offers the possibility of creating artificial experiences in real time, that make the user feel immersed and able to interact as if it was the real world. Additionally, virtual reality therapy allows for personalization of the therapy to match the specific social challenges of each patient.

Preliminary findings suggest virtual reality exposure to lead to faster symptom reduction than traditional therapy and may therefore be cost-effective. While the potential beneficial effects of virtual reality exposure to challenging social situations, that taps social cognitive functions, are evident and virtual reality therapies are promising in general, the research field is in urgent need of evidence on the effectiveness of virtual reality therapy in adults with ASD.

The STEPS trial evaluates the effect of a Virtual Reality-based pro-functional, Social Cognitive Training (VRSCT) versus treatment as usual. We expect to find VRSCT to be more beneficial in improving social cognitive deficits, daily life functioning, and quality of life in adults with ASD.

If the results of the current trial are positive, this short-term, manualised treatment using well-tested VR-software, can easily be implemented in clinical practice, that is in the psychiatric out-patient facilities or in community-based facilities where it can benefit a large group of suffering ASD patients. Additionally, it can be adapted for use in related clinical target groups such as adolescents with ASD or patients with psychosis experiencing social cognitive and functional deficits.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 years or older
2. Ability to give informed consent
3. Diagnosis of an autism spectrum disorder (ICD-10 code F84.0; F84.1; F84.5; F84.8)
4. T-score on SRS-A self-report ≥ 60

Exclusion Criteria:

1. Rejecting informed consent
2. A diagnosis of organic brain disease
3. Intellectual disability (IQ ˂ 70)
4. A command of spoken Danish or English inadequate for engaging in therapy
5. ADHD-diagnosis with untreated symptoms
6. Displaying an imminent homicidal or suicidal risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Social Responsiveness Scale, Adult Version, Self-report | Baseline, 3 month follow-up and 6 month follow-up
  The primary outcome is level of social impairment is measured by the Social Responsiveness Scale, Second Edition, Adult version, Self-report (SRS-2A) at cessation of treatment at 3-months.
  SRS-2A measures the presence and severity of social impairment in everyday life. The SRS-2A is a commonly used measure in autism spectrum research and has demonstrated good reliability and validity.
  SRS-2A is a 65-item rating scale, scored on on a 4-point Likert Scale (0-3). Each item is scaled from 0 (never true) to 3 (almost always true), generating a total score ranging from 0 to 195. The SRS-2A is provides a continuous measure of social impairment, where a higher score reflects a greater degree of difficulties with social interactions in everyday life.
  Follow-up assessments will comprise ratings of the previous two-week period.

SECONDARY OUTCOMES:
Social Responsiveness Scale, Adult Version, Informant Report | Baseline, 3 month follow-up and 6 month follow-up
  Social Responsiveness Scale, Adult Version, Informant Report is a 65-item rating scale, scored on on a 4-point Likert Scale (0-3). Each item is scaled from 0 (never true) to 3 (almost always true), generating a total score ranging from 0 to 195. The SRS-2A is provides a continuous measure of social impairment, where a higher score reflects a greater degree of difficulties with social interactions in everyday life. Follow-up assessments will comprise ratings of the previous two-week period.
Social Interaction Anxiety Scale (SIAS) | Baseline, 3 month follow-up and 6 month follow-up
  SIAS is a self-report questionnaire measuring social anxiety in social interaction. SIAS consists of 20 items that are rated on a 5-point Likert scale ranging from 0 (not at all characteristic of me) to 4 (extremely characteristic of me). Item 5, 9 and 11 are positively worded items and have reverse scoring. A total SIAS score is generated by summing the ratings ranging from 0 to 80. Higher scores reflects a higher degree of social anxiety in social interaction.
The Empathy Quotient | Baseline, 3 month follow-up and 6 month follow-up
  The Empathy Quotient (EQ) is a 60-item questionnaire designed to measure empathy in adults. Each item is scored on a 4-point scale (strongly agree, slightly agree, slightly disagree, strongly disagree).
  Items 1, 6, 19, 22, 25, 26, 35, 36, 37, 38, 41, 42, 43, 44, 52, 54, 55, 57, 58, 59, and 60 are assigned two points if rated as 'strongly agree' and one point if rated 'slightly agree.'
  Items 4, 8, 10, 11, 12, 14, 15, 18, 21, 27, 28, 29, 32, 34, 39, 46, 48, 49, and 50 are assigned two points if rated as 'strongly disagree' and one point if rated 'slightly disagree.'
  The minimum score achievable is 0, and the maximum score is 80. A higher score indicates higher levels of empathy in adults.
The High Risk Social Challenge Task (HiSoC) | Baseline, 3 month follow-up and 6 month follow-up
  The High Risk Social Challenge task (HiSoC) is a standardized, performance-based task assessing social skills in terms of affect, odd behaviour and language and social-interpersonal skills. Following a short verbal instruction, the participants are being video-taped for 45 seconds while performing a task.
  HiSoC consists of 16 items that are rated on a 5-point Likert scale from 1 to 5. Smaller ratings reflect low levels of appropriate, effective social behavior. Larger ratings reflect high levels of appropriate, effective social behavior. A total HiSoC score is generated by summing the rating ranging from 16 to 80. Higher scores reflects a higher degree of social skills.
Emotion Recognition Task (CANTAB ERT) | Baseline, 3 month follow-up and 6 month follow-up
  Computer-morphed images derived from the facial features of real individuals, each showing a specific emotion, are displayed on the screen, one at a time. Each face is displayed for 200ms and then immediately covered up to prevent residual processing of the image. The participant must select which emotion the face displayed from 6 options (sadness, happiness, fear, anger, disgust or surprise).The outcome measures for ERT cover percentage and number correct or incorrect and overall response latencies, which can be looked at either across individual emotions or across all emotions at once.

OTHER OUTCOMES:
CAT-Q (Camouflaging Autistic Traits Questionnaire) | Baseline, 3 month follow-up and 6 month follow-up
  The Camouflaging Autistic Traits Questionnaire (CAT-Q) is a 25-item self-report measure of social camouflaging behaviours for individuals of age 16 and above. Each item is rated on a likert scale from 1 (Strongly Disagree) to 7 (Strongly Agree). The total score ranges from 25-175 with higher scores reflecting greater degree of camouflaging.
SR-AS (Questionnaire on sensory reactions) | Baseline, 3 month follow-up and 6 month follow-up
  The SR-AS is a self-report instrument for sensory reactivity. It can be used for evaluation of sensory symptoms as described in DSM-5 for autism spectrum conditions. The instrument comprises statements about reactions to sensory input. The task is to self-rate the statements rated on a likert scale from 0 (Totally Disagree) to 3 (Totally Agree). Total scores ranges from 0 - 96.
Beck Depression Inventory (BDI) | Baseline, 3 month follow-up and 6 month follow-up
  The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. Each item is rated on a 4-point scale from 0 (symptom absent) to 3 (severe symptoms). The total score ranges from 0 to 63, with higher scores reflecting greater degree of depressive symptoms.
Intolerance of Uncertainty Scale (IUS-12) | Baseline, 3 month follow-up and 6 month follow-up
  The Intolerance of Uncertainty Scale (IUS-12) is a 12-item, self-report questionnaire measuring the tendency to think or react negatively toward uncertain events. IUS-12 consists of 12 items (e.g., "It frustrates me not having all the information I need") and is scored on a 5-point Likert scale from 1 ("Not at all characteristic of me") to 5 ("Very Characteristic of me"). The total score ranges from 12 to 60. A greater score indicates a greater level of negative reactions towards uncertainty.
General Alexithymia Factor Score (GAFS-8) | Baseline, 3 month follow-up and 6 month follow-up
  The General Alexithymia Factor Score (GAFS-8) is a 8-item, self-administered questionnaire that measures alexithymia.
  Each item is scored on a 5-point Likert-type scale 1 (strongly disagree) to 5 (strongly agree). Total score is ranging from 8 to 4, with higher scores indicating greater impairment/challenges.
The Repetitive Behaviour Questionnaire-3 (RBQ-3) | Baseline, 3 month follow-up and 6 month follow-up
  RBQ-3 is a 20-item self-report questionnaire that measures of restricted and repetitive behaviours and interests (RRBIs). All items are scored on a 4-point Likert-type scale ranging from 1 (Never or rarely) to 5 (30 or more times daily/Serious or extreme/Serious or severe).
  RBQ-3 Mean Total Score is obtained adding each individual's score of 1, 2, 3 or 4 across every item in the questionnaire. This total is then divided by the number of items completed for each individual. A score of between1-4 is generated. A higher mean score reflects higher level of RRBIS.
Inventory of Psychotic-Like Anomalous Self-Experiences (IPASE) | Baseline, 3 month follow-up and 6 month follow-up
  Inventory of Psychotic-Like Anomalous Self-Experiences (IPASE) is a self-report measure of minimal self-disturbance. IPASE consists of 57-item self-report scale in which participants indicate how much they agree with statements on a scale ranging from 1 (strongly disagree) to 5 (strongly agree). Total score ranges from 57 to 285. Higher scores reflects more psychotic-like anomalous self-experiences.
Green Paranoid Thought Scale (GPTS) | Baseline, 3 month follow-up and 6 month follow-up
  The Green Paranoid Thought Scale consists of a 32 item self-report measure of paranoia designed for both clinical and non-clinical populations.
  Part A assesses ideas of reference (e.g. 'It was hard to stop thinking about people talking about me behind my back') and Part B assesses ideas of persecution (e.g. 'I was convinced there was a conspiracy against me').
  Each item is rated on a five-point scale (1-5). Scores on each scale can range from 16 to 80. Higher scores indicate greater levels of paranoid thinking.
Adult ADHD Self-Report Scale (ASRS) | Baseline, 3 month follow-up and 6 month follow-up
  The Adult ADHD Self-Report Scale (ASRS) is an 18-item self-report questionnaire designed to assess Attention Deficit Hyperactivity Disorder (ADHD) symptoms in adults.
  The ASRS consists of an 18-item scale evaluating the dimensions of inattention and hyperactivity-impulsiveness subtypes of ADHD in adults.
  The ASRS full edition consists of nine items that represent symptoms related to inattention (items 1-4 and 7-11), and nine items assessing symptoms of hyperactivity-impulsiveness (items 5-6 and 12-18). Each of the items is scored on a five-point Likert rating scale with 0="never", 1="rarely", 2="sometimes", 3="often", and 4="very often" based on the participant's experiences over the last 6 months. A high score indicates a greater severity of self-reported ADHD symptoms.
  Assessments will comprise ratings of the previous 1-month period.
Social Skills Performance Assessment (SSPA) | Baseline, 3 month follow-up and 6 month follow-up
  The SSPA is a performance-based test, that measure social behaviour. SSPA consists of two communication scenarios: One that involves the participants introducing themselves to a new neighbour and one that involves the participants requesting their landlord to fix a leak after the landlord had previously agreed to fix the leak but had never completed the task.
  The test is measuring both social competence and appropriateness and is scored on 17 items in total.
  All items are rated on a five-point (1-5) scale, with 1 as the lowest and 5 as the highest score.
  In scenario one the minimum score is 1*8=8. The maximum score: 5*8=40.
  In scenario two, the minimum score: 1*9=9. Maximum score: 5*9=45.
  The SSPA Total score ranges from 17 to 85. Higher scores reflect higher social competence and appropriateness.
WHO-5 Well-Being Index (WHO-5) | Baseline, 3 month follow-up and 6 month follow-up
  WHO-5 is a self-report questionnaire assessing subjective psychological well-being. The questionnaire consists of 5 items and is scored from 0 (At no time) to 5 (all of the time).
  The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
General Self Efficacy Scale (GSE) | Baseline, 3 month follow-up and 6 month follow-up
  GSE is a self-report questionnaire assessing perceived self-efficacy. GSE consists of 10 items rated on a Likert scale ranging from 1 (not at all true) to 4 (exactly true). Higher scores indicate greater self-efficacy. Total score ranges from 10 to 40.
EuroQOL five dimensions questionnaire (EQ-5D) | Baseline, 3 month follow-up and 6 month follow-up
  EQ-5D is a self-report questionnaire measuring health-related quality of life. The questionnaire is a description of the subject's current health in 5 dimensions i.e., mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The subject is asked to grade their own current level of function in each dimension into one of three degrees of disability (severe, moderate or none). The combination of these with the conditions "death" and "unconscious" enables description of 245 different health states.
  The EQ-5D will be used for health outcomes studies and economic analyses
Defeatist Performance Attitude Scale (DPAS) | Baseline, 3 month follow-up and 6 month follow-up
  DPAS contains 15 items assessing an individual's tendency to overgeneralize from past failures to expected future failures (e.g. "If I fail partly, it is as bad as being a complete failure", "People will probably think less of me if I make a mistake", "If I ask a question, it makes me look inferior"). Scoring for these items is on a 7 point scale (1-7) with higher scores indicating greater severity of defeatist attitudes (range for DPAS total = 15-105).
Temple University Community Participation Measure (TUCP) | Baseline, 3 month follow-up and 6 month follow-up
  TUCP is a self-report questionnaire measuring participation in community activities during the last 30 days.
  TUCP assess 26 areas of life, such as working for pay, going to a movie and going to a library with 26 items.
Personal and Social Performance Scale (PSP) | Baseline, 3 month follow-up and 6 month follow-up
  PSP is a a semi-structured interview assessing daily life social functioning in the domains social relations, job/education, personal hygiene, aggressive behaviour.
  Scores ranging from 1-100, with a score of 100 reflecting the best personal and social functioning
Davos Assessment of the Cognitive Biases Scale (DACOBS) | Baseline, 3 month follow-up and 6 month follow-up
  DACOBS is a self-report questionnaire measuring cognitive biases. 42 Items are rated on a 7-point Likert scale, ranging from 1 (Strongly disagree) to 7 (Strongly agree) with higher scores indicating more strongly held cognitive biases.
  Total scores ranging from 42-294.
The Awareness of Social Inference Test - Short Form, part 2 Social Inference, Minimal (TASIT-S) | Baseline, 3 month follow-up and 6 month follow-up
  The TASIT-S is a measure of emotion perception and Theory of Mind.
  The TASIT-S part 2 Social Inference - Minimal is a Theory of Mind task, that is comprised of 9 video clips depicting sincere (4 items) and sarcastic interactions (5items) between two actors.
  For each video 4-items is scored. Total scores ranging from 4*0 = 0 to 4*9=36.
The Hinting Task | Baseline, 3 month follow-up and 6 month follow-up
  The Hinting task measures ability to infer others' true intentions from indirect speech. Participants read 10 vignettes of two characters interacting, ending with one character hinting at his or her true thoughts, feelings, or intentions. Participants give open-ended responses of what the character truly meant, and if their answer is wrong, the experimenter reads a second hint. Answering correctly on the first hint yields two points, while the second hint yields one. The hinting task is scored for total correct out of 20. Minimum score is 0 and maximum score is 20.
Behavior Rating Inventory of Executive Function - Adult Version, Self-Report (BRIEF-A, Self-Report) | Baseline, 3 month follow-up and 6 month follow-up
  BRIEF-A is a self-report questionnaire, that includes 75 items assessing executive function. Participants rate whether a specific behavior is a problem on a 3-point Likert scale (0 = Never, 1 = Sometimes, 2 = Often). The global score (General Executive Function) ranges from 0-225. Higher scores indicate more problems with executive functioning.
Client Satisfaction Questionnaire (CSQ) | 3 month follow-up
  CSQ is an 8 item self-report measuring client satisfaction with the intervention. All items are scored on a 4-point Likert scale ranging from bad (1) to excellent (4). Higher scores indicate higher satisfaction.
Negative Effects Questionnaire (NEQ) | 3 month follow-up
  NEQ is a 32-item self-report questionnaire measuring negative events and outcomes in the participants life during the intervention period.
  All items are rated on a 5-point Likert scale ranging from 0 (not at all) to 4 (very much). Higher score reflects higher rate of negative events.
Multimodal Presence Scale, Modified Shortened Danish Version (MPS-MSDV) | 3 and 10 weeks post baseline
  MPS-MSDV is a self-report questionnaire measuring presence in virtual reality. The modified, shortened Danish Version consist of 10 selected items scored on a 5-point Likert Scale ranging from 1 (Strongly disagree) to 5 (Strongly agree). Higher scores reflect higher degree of presence in Virtual Reality. The MPS-MSDV will be administered only to participants in the experimental group.
Virtual Reality Simulation Sickness Questionnaire, Modified Danish Version (VRSSQ-MDV) | 3 and 10 weeks post baseline
  VRSSQ-MDV is a is a self-report questionnaire measuring virtual reality simulation sickness. The Modified Danish Version consist of 9 items rated on a 4-point Likert Scale ranging from 0 (not at all) to 3 (a lot). Higher scores reflect higher degree of virtual reality simulation sickness. The VRSSQ-MDV will be administered only to participants in the experimental group.
Readiness for Therapy Questionnaire (RTQ) | 1 week post baseline
  RTQ is a 6-item self-report questionnaire measuring the participants positive attitude and preparedness to enter therapy for the purpose of resolving problems. Each item is scored on a 5-point Likert scale ranging from strongly disagree (0) to strongly agree (4). Item 2, 3 and 6 are reversed scored. A higher score indicated greater readiness for therapy. The RTQ will be administered only to participants in the experimental group.

CONTACTS AND LOCATIONS:
Overall Officials: Louise B. Glenthøj, DrMSc, Principal Investigator — Copenhagen Research Centre for Mental Health (CORE), Mental Health Centre Copenhagen
Locations (1):
- Copenhagen Research Centre for Mental Health (CORE), Mental Health Centre Copenhagen, Mental Health Services in the Capital Region, Denmark, Copenhagen, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No